CLINICAL TRIAL: NCT06334770
Title: Influence of Roxolid Implant Material on the Implant Stability of Maxillary Implant Retained Overdenture
Brief Title: Influence of Roxolid Implant Material on the Implant Stability Implant Stability
Acronym: BLX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amany Ibrahim, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASuRecD032136
Record Dates: First submitted 2024-03-20; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Completely Edentulous Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group( A) ROXOLID IMPLANT (Experimental): NINE patients were rehabilitated with implant retained maxillary overdenture where four Straumann BLX® ROXOLID implant were inserted opposed by mandibular complete denture.
  Interventions: Device: Roxolid implants
- Group (B) CONVENTIONAL TITANIUM IMPLANT (Active Comparator): NINE patients were rehabilitated with implant retained maxillary overdenture where four conventional titanium implants were inserted opposed by mandibular complete denture.
  Interventions: Device: Titanium implants

INTERVENTIONS:
Device: Roxolid implants — four Straumann BLX® roxolid implant 15% zirconium and 85% titanium), 3.7 mm in diameter, and 10 mm in length.implants were selected with the following criteria: tapered, self-tapping, aggressively threaded,were inserted with novalock attachments.
  Other Names: Straumann BLX® SLA implants
  Arms: Group( A) ROXOLID IMPLANT
Device: Titanium implants — four conventional acid etched pure implants tapered, self-tapping, threaded, two-piece, with the 10 mm length and 3.7 mm diameter were inserted with Sphero flex attachments.
  Other Names: JD EVOLUTION PLUS implants
  Arms: Group (B) CONVENTIONAL TITANIUM IMPLANT

SUMMARY:
Fourteen completely edentulous patients were selected to participate in this study. From the outpatient clinic of Prosthodontic Department, Faculty of Dentistry, Ain Shams University.

After fabrication of complete denture for all patients, patients were randomly divided to:

Group A: Seven patients were rehabilitated with implant retained maxillary overdenture where four Straumann BLX® implant were inserted opposed by mandibular complete denture.

Group B: Seven patients were rehabilitated with implant retained maxillary overdenture where four conventional acid etched implants were inserted opposed by mandibular complete denture.

After implant placement using surgical guide, smart peg and ostell device were used to measure the primary stability of the implant then cover screw was placed and after six weeks, secondary stability was measured for both groups.

After four months, the second stage started in which exposure of the implant fixtures took place and pick up was carried out.

Patients were recalled frequently for post-insertion inspection and adjustment.

DETAILED DESCRIPTION:
Background: long term success of implant restoration depends on many factors one of them is the sufficient implant stability which is lowered in compromised bone density sites such as the maxilla which is categorized as type III & IV bone, so searching for new innovation and updates in implant material and features is very mandatory. So, the aim of this study was asses and compare between two implant materials roxolid versus traditional titanium on the primary and secondary stability.

Methods: eighteen completely edentulous patients were selected they all received maxillary implant retained overdentures and lower complete dentures, they were divided equally in to two groups according to the type of the material of the implants. Group A received a total number of 36 (Roxolid) Implants were made of roxolid material and Group B received a total number 36 (Titanium) implants were made of traditional titanium alloys. Implant stability was assed using ostell device, the primary implant stability was measured at the day of implant installation however, secondary implant stability was measured after six weeks of implant placement. Paired t-test was used to compare between primary and secondary stability in the same group and independent t-test was used to compare between the two groups with a significant level < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients as the last extraction should be at least six months before implant placement.

  * Patients with good oral hygiene.
  * Sufficient inter arch space (11 mm) which were diagnosed by mounted diagnostic casts.
  * Firm and healthy mucosa covering the residual alveolar ridge.

Exclusion Criteria:

* - Heavy smokers.
* Patients with para functional habits.
* Patients had TMJ disorders.
* Patients had systemic disease that could interfere with implant placement or affect bone healing such as; thyroid and uncontrolled diabetes.
* Patients undergoing chemo and radiotherapy.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
measuring primary at time of surgery | same day of implant placement
  using an Ostell device with a smart peg to measure primary stability at the time of implant placement and measuring secondary stability after six weeks of implant placement.

SECONDARY OUTCOMES:
secondary implant stability after 6 weeks | 6 weeks
  measuring secondary stability using ostell device and smart peg

CONTACTS AND LOCATIONS:
Overall Officials: shaimaa L mohamed, PROFESSOR, Principal Investigator — Ains hams univeristy
Locations (1):
- Faculty of Dentistry of Dentistry Ainshams Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
THE PROTOCOL OF OUR STUDY THAT WILL BE SHARED
Supporting Information: Study Protocol
Time Frame: The data is already available
Access Criteria: A link contains the pdf of the study protocol
URL: https://drive.google.com/file/d/1UGyxP3rqdopNavtuEMN79s6cwtl2I57f/view?usp=sharing

REFERENCES:
- [Background] Pandey C, Rokaya D, Bhattarai BP. Contemporary Concepts in Osseointegration of Dental Implants: A Review. Biomed Res Int. 2022 Jun 14;2022:6170452. doi: 10.1155/2022/6170452. eCollection 2022. PMID 35747499
- [Background] Thanasrisuebwong P, Pimkhaokham A, Jirajariyavej B, Bencharit S. Influence of the Residual Ridge Widths and Implant Thread Designs on Implant Positioning Using Static Implant Guided Surgery. J Prosthodont. 2023 Apr;32(4):340-346. doi: 10.1111/jopr.13557. Epub 2022 Jun 22. PMID 35686699
- [Derived] El-Hady AIA, Eid HI, Mohamed SL, Fadl SM. Influence of titanium and titanium-zirconium alloy as implant materials on implant stability of maxillary implant retained overdenture: a randomized clinical trial. BMC Oral Health. 2024 Aug 6;24(1):902. doi: 10.1186/s12903-024-04692-x. PMID 39107737